CLINICAL TRIAL: NCT03696420
Title: Probabilistic Determination of the Ventro-intermediate Nucleus of the Thalamus (VIM) Coordinates From Radio-anatomical Landmarks on 1.5 Tesla MRI
Brief Title: Probabilistic Targeting of the VIM
Acronym: PROBA-VIM
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de Recherche en Informatique et en Automatique (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/26
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Essential Tremor; Deep Brain Stimulation
Keywords: Probabilistic targeting; VIM-DBS; Machine-learning; Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DBS surgery targeting the VIM: Patient who underwent a DBS surgery targeting the VIM at Bordeaux University Hospital
  Interventions: Other: Coordinates of active plots and VIM landmarks calculation

INTERVENTIONS:
Other: Coordinates of active plots and VIM landmarks calculation — Stimulation efficacy will be assessed by comparing, according to usual care, the clinical evaluation (FTM scale) with and without stimulation, and the four contacts of each electrode will be tested clinically, with an accelerometer and an electromyography to determine which one is the most active on tremor. Coordinates of the anatomical landmarks will be calculated on the pre-operative MRI and those of the active plots on the fusion between post-operative CT-scan and pre-operative MRI.

SUMMARY:
After having included the most improved patients by DBS among those implanted in Bordeaux Hospital University, and having defined the most active plots on tremor by its prospective grading on Fahn-Tolosa-Marin (FTM) scale and accelerometry, coordinates of active plots and landmarks will be calculated on post-operative imaging. Association between landmarks and active plots coordinates will be modelled with machine-learning algorithms. The aim is to retrieve the position of the VIM on the basis of the landmarks coordinates.

DETAILED DESCRIPTION:
The intermedius ventralis nucleus of the thalamus (VIM), which represents the target for deep brain stimulation (DBS) in essential tremor, still remains invisible to imaging in spite of the development of new MR sequences. The coordinates currently used in the classical (ACPC) system are so imprecise that per-operative electrophysiology is mandatory to locate the exact position of this target. Micro-electrode recordings (MER) however improve hemorrhagic risk and may be poorly tolerated by patients operated on 7 to 8 hours under local anaesthesia. Based on litterature review, no one tried to retrieve the position of the VIM from anatomical landmarks coordinates in the era of MRI. The patients operated will be clinically tested to define those very well improved by the stimulation. Stimulation efficacy will be assessed by comparing the clinical evaluation (FTM scale) with and without stimulation, and the four contacts of each electrode will be tested clinically, with an accelerometer and an electromyography to determine which one is the most active on tremor. Coordinates of the anatomical landmarks will be calculated on the pre-operative MRI and those of the active plots on the fusion between post-operative CT-scan and pre-operative MRI. These coordinates will be analysed by machine-learning algorithms to create a model predicting the position of the active contacts from the coordinates of the landmarks.

ELIGIBILITY:
Inclusion Criteria:

* patient older than 18 years
* who underwent a DBS surgery targeting the VIM at Bordeaux University Hospital
* in the strict indication of the essential tremor
* with an excellent post-operative result defined by a complete withdrawal of medication, a stability of the stimulation effects without any setting adjustments since at least 3 months and an improvement of more than 66% on the FTM scale between OFF and ON-stimulation assessments.

Exclusion Criteria:

- patients who underwent a DBS surgery targeting the VIM for different indications (Parkinson's disease for instance), patients with a poor post-operative efficacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who underwent a DBS surgery targeting the VIM at Bordeaux University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Euclidian distance between the predicted target and the center of the active contact of the DBS lead | 6 month after DBS surgery
  Euclidian distance in milimeter measured on the fusion between post-operative CT-scan and pre-operative MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Nejib ZEMZEMI, MD-PhD, Study Chair — Institut National de Recherche en Informatique et en Automatique
Locations (1):
- Bordeaux University Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No